CLINICAL TRIAL: NCT05868109
Title: Inhaled Nitric Oxide for Cardiac Arrest in Pediatrics and Adults (iNOCAPA): A Pilot Randomized Controlled Trial and Translational Biology Study
Brief Title: Inhaled Nitric Oxide for Cardiac Arrest in Pediatrics and Adults (iNOCAPA)
Acronym: iNOCAPA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other)
Responsible Party: Principal Investigator, Jamie Hutchison, Principal Investigator, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1822
Record Dates: First submitted 2022-12-01; First posted 2023-05-22 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Cardiac Arrest
Keywords: Neuroprotection; Nitric Oxide
MeSH Terms: conditions — Heart Arrest | interventions — Endothelium-Dependent Relaxing Factors; salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The nitric oxide delivery device is covered with a secure shroud and Respiratory Therapists (RTs) are able to safely administer the nitric oxide or sham and document nitric oxide dose and their delivery device checks and monitor for adverse effects according to there clinical standard of care throughout the study intervention. The RTs also document whether there has been a unmasking of the intervention every 12 hours.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants with Sham (no nitric oxide) (Sham Comparator): The mechanical ventilator circuit of the study participants are attached to the inhaled nitric oxide delivery device but nitric oxide is not delivered.
  Interventions: Drug: Sham
- Participants with Nitric Oxide (Experimental): The mechanical ventilator circuit of the study participants are attached to the inhaled nitric oxide delivery device and nitric oxide is delivered.
  Interventions: Drug: inhaled nitric oxide (iNO)

INTERVENTIONS:
Drug: inhaled nitric oxide (iNO) — In patients randomized to the this arm, iNO will be delivered into the ventilator circuit through the endotracheal tube or tracheostomy. The dose will be 80 ppm during chest compressions and reduced to 20 ppm immediately following ROC. If the patient is enrolled following ROC, the dose will be 20 ppm. Dose modifications will occur if there is toxicity or if there is a clinical concern. The iNO or sham will be continued for 72 hours or until extubation.
  Other Names: INOMAX
  Arms: Participants with Nitric Oxide
Drug: Sham — In patients randomized to sham, the iNO delivery device will be connected to the ventilator circuit or manual ventilation bag but flow of iNO will not be turned on. For the purposes of patient safety and to maintain blinding, the respiratory therapists (RTs) will continue checks of gas flow, flow adjustments and change iNO gas tanks at rates like routine clinical procedures on patients treated with iNO or sham.
  Other Names: Sham intervention with no flow of inhaled nitric oxide to the patient
  Arms: Participants with Sham (no nitric oxide)

SUMMARY:
This study is a multi-center, double blind, randomized controlled trial of inhaled nitric oxide (iNO) in children and adults with cardiac arrest (CA). The purpose of this pilot study is to test the feasibility of rapidly randomizing patients to iNO or sham treatment during cardiopulmonary resuscitation (CPR) or shortly after return of circulation (ROC) and evaluate blood biomarkers associated with iNO compared to sham. Return of circulation may refer to return of spontaneous circulation (ROSC) or ROC through extracorporeal cardiopulmonary resuscitation (E-CPR).

DETAILED DESCRIPTION:
Background: Sudden cardiac arrest is a leading cause of death and neurological handicaps but there is no neuroprotective drug which improves outcome. Recently we discovered a blood biomarker of response to a neuroprotective therapy in our pre-clinical model of cerebral ischemia-reperfusion injury. Biomarkers will likely be used, in the future, to assess response to specific neuroprotective drugs and to help titrate drug dose and duration in individual patients.

Inhaled nitric oxide (iNO) has recently been shown to improve return of spontaneous circulation, survival, and neurological outcome in animal models of cardiac arrest. We have therefore started a pilot randomized controlled trial (RCT) and translational biology study of iNO in children and adults with cardiac arrest. This study will help us design future fully powered RCTs of iNO. We will use methods, from our pre-clinical model, to discover blood biomarkers of response to therapy.

Objectives: In patients with cardiac arrest: (1) Test the safety and feasibility of rapidly randomizing patients to iNO or sham during chest compressions, or shortly after return of circulation (ROC), either spontaneous or by extracorporeal life support. (2) Maintain blinding and measure study outcomes for 6 months post-arrest. (3) Use immunoassays, mass spectrometry and fluorometric assays to determine the differences in serum protein, nitrite, and nitrate biomarker concentrations between the two intervention groups and discover blood biomarkers of therapeutic response to iNO.

Patient population and sample size: Pediatric and adult (total N=40) patients with cardiac arrest admitted to 8 intensive care units (ICUs) at 4 hospitals: SickKids, University Health Network - Toronto General Hospital (TGH) and Toronto Western Hospital (TWH) and Unity Health - St. Michael's Hospital (SMH).

Methods: All patients meeting eligibility criteria will be enrolled, during chest compressions or within 6 hours of ROC, using deferred consent. Patients will be randomized to iNO or sham procedures, using a Redcap screening and randomization tool. Registered respiratory therapists will rapidly start the study gas using our blinded study apparatus. Inhaled NO will be started at a dose of 80 ppm via the endotracheal or tracheostomy tube during chest compressions and reduced to, or started at, 20 ppm after ROC. The iNO or sham procedures will be continued for 72 hours, and weaned off over 12 hours, or stopped earlier if the patient is extubated or dies. Using the Utstein data template for cardiac arrest research, we will collect data into an electronic case report form and Oracle database. Survival, cerebral performance category scores and quality of life scores will be assessed at 1 and 6 months following cardiac arrest. Data and documentation will be reviewed intermittently to ensure that we are compliant with Health Canada guidelines for drug trials.

Serum is being collected and banked at 4 time points following cardiac arrest. The concentrations of biomarkers will be measured and compared between the 2 intervention groups.

Progress: This study is funded by the Heart and Stroke Foundation of Canada.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in this study, an individual must meet all the following criteria:

1. Aged 1 day* to 80 years on the day the study intervention is started
2. In-hospital or out-of-hospital CA with CPR > 5 minutes
3. It is possible to randomize and start the iNO or sham during CPR or within 5 hours of ROC**
4. Mechanically ventilated in a study site ICU

Note: *Age 1 day is defined as 24 hours and a minimum corrected gestational age ≥ 38 weeks.

Note: **ROC refers to either ROSC or ROC via extracorporeal cardiopulmonary resuscitation (E-CPR).

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Unwitnessed cardiac arrest
2. Cardiac arrest due to birth asphyxia
3. Pre-arrest poor neurologic function*
4. Already receiving iNO at the time of CA
5. Any condition or diagnosis, in the opinion of the PI, Co-Investigators, or MRPs, in which iNO would have adverse effects on physiology or where the cardiac anatomy and physiology has not yet been adequately assessed
6. Any condition or diagnosis, in the opinion of the PI, Co-Investigators, or MRPs, in which iNO would be indicated as therapy post-arrest
7. CPR duration > 45 minutes; if less than 18 years old, in-hospital CPR duration > 60 minutes**
8. Known pregnancy***
9. Terminal illness ʈ

Note: * Poor neurologic function is defined as CPC ≥ 4 or PCPC ≥ 4.

Note: **CPR duration is defined as total cumulative duration of CPR (i.e., if a patient has multiple arrests with CPR, the duration of these will be added); patients who undergo E-CPR will not be excluded, to maximize recruitment for this feasibility trial.

Note: ***B-HCG screening is not required for enrollment in women of reproductive age, but testing will occur as soon as possible (within 6 hours of enrollment).

Patients who are cannulated to ECMO for cardiorespiratory support will NOT be excluded a priori.

ʈ The MRP knew that the patient was dying pre-arrest

Ages: 1 Day to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-08-31 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Drug Procedural Feasibility | We will monitor screening numbers, rates of enrolment of eligible patients and delivery of study intervention according to CONSORT criteria over the 2 year timeframe of study enrolment.
  Number of successful initiations of iNO or sham among the 40 patients enrolled in the study. We will monitor and improve our rates of enrolment and study intervention by examining and improving upon factors related to protocol compliance.
Drug Procedural Feasibility | We will monitor compliance to the study intervention during the 72 hours of drug/sham delivery and 12 hours of weaning and stopping the study intervention on each enrolled patient over the 2 years of study enrolment.
  Number of successful continuations of iNO or sham for 72 hours followed by weaning and stopping the study intervention over the next 12 hours. Using real time monitoring of the study intervention we will optimize compliance to the full duration of the study intervention and improve upon any deviations to the study intervention over the full 72 + 12 hours of the study protocol.

SECONDARY OUTCOMES:
Monitor recruitment rate | For study duration, approximately 2 years.
  Recruitment rate is the rate of enrolment/randomization/consent divided by the number of eligible patients which meet all inclusion criteria and have no exclusion criteria.
Monitor time to randomization of eligible patients | At study enrollment during the 2 years of study recruitment.
  Timing of randomization. The time of randomization following onset of cardiac arrest will be recorded. We will attempt to speed up this time using simulations with study and clinical personnel and by debriefing each enrolled patient with the teams involved. We will attempt to enrol some patients who have a cardiac arrest in the ICU during chest compressions and for those patients enrolled following return of circulation, the timeframe is a maximum of 5 hours.
Monitor masking and unmasking events | During the 2 year study duration and data analysis.
  Number of unblinding instances. The study apparatus (inhaled nitric oxide gas delivery device) has a secure cover that only the Respiratory Therapists are trained to open. The RTs will record any unblinding events which may include breaking/cutting of the cover ties and opening of the apparatus cover by clinical personnel other than RTs. The RTs will record and sign 'unblinding yes/no' into their masked RT study case report form on each RT clinical shift and study Research Coordinators will enter this data into the study electronic database. We will monitor unblinding events in real time and attempt to prevent these from happening.
Study follow-up rates | For study follow-up, approximately 2.5 years.
  We will measure outcomes at 1 and 6 months following cardiac arrest as outlined in more detail below. Number of completed study outcomes at 6 months following cardiac arrest will be followed in real time and we will attempt to maximize follow-up rates.

OTHER OUTCOMES:
Return of spontaneous circulation (ROSC) | Duration of study enrollment, approximately 2 years.
  Rate of ROSC, for participants in whom the iNO or sham procedure is initiated during chest compressions and cardiopulmonary resuscitation.
Survival at hospital discharge | For duration of study follow-up, approximately 2 years and 6 months.
  Survival to hospital discharge, 1 month, and 6 months following cardiac arrest.
Cerebral performance category score | For duration of study follow-up, approximately 2 years and 6 months.
  Cerebral Performance Category (CPC) or Pediatric Cerebral Performance Category (PCPC) scores, for adults and children respectively, at 1 month, and 6 months following cardiac arrest. CPC scores range from 1 to 5 with 1 indicating good outcome, 4 indicating persistent vegetative state and 5 indicating death. PCPC scores range from 1 to 6, with 1 indicating good cerebral performance, 5 indicating persistent vegetative state and 6 indicating death.
Quality of Life Score | For duration of study follow-up, approximately 2 years and 6 months.
  Pediatric Quality of Life (PedsQL) scores (includes 2 adult versions) at 1 month, and 6 months following cardiac arrest. Results are reverse scored and transformed into a scale with a range of 0 to 100, with higher scores indicate better health related quality of life.
Quality of life after brain injury | For duration of study follow-up, approximately 2 years and 6 months.
  Quality Of Life after Brain Injury-Overall Scale (QOLIBRI-OS, for adults only) at 1 month, and 6 months following cardiac arrest. QOLIBRI scores are reported on a 0 to 100 scale, with 0 indicating worst possible quality of life and 100 indicating best possible quality of life.
Blood protein biomarkers | Bloods sampled and banked for up to 7 days post-cardiac arrest. Biomarker measurements will be done after we have recruited 40 patients into the study. i.e. at approximately 2 years after the start of study enrolment.
  Blood will be sampled, and the serum separated and divided into aliquots and banked at 4 time points following enrolment. These time points are within 4 hours following enrolment and with AM clinical blood sampling on Day 2, 4 and 7. Day 1 is defined as the 24 hour period from 00:01 to 24:00 hours during which the patient was enrolled. At the end of the study, a panel of brain specific and inflammatory proteins will be measured in serum samples and their concentrations compared between intervention groups. We will also perform shotgun proteomics using untargeted mass spectrometry and compare blood peptide/protein concentrations from Day 2 samples between the 2 intervention groups. Promising peptides/proteins that may indicate response to iNO will then be measured, using targeted mass spectrometry in serum samples from all 4 time points to determine the time course of these peptides/proteins.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Hutchison, MD, Principal Investigator — The Hospital for Sick Children
Locations (4):
- Canada (4):
  - St. Michael's Hospital, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - The Hospital for Sick Children, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
All de-identified individual participant data (IPD) that underlie results in a publication will be shared upon request. The study protocol, and statistical analysis plan will be shared starting 6 months after publication upon request in writing.
  Requests for IPD will be reviewed by the study PI and SickKids institute. IPD will be provided to researchers interested in furthering academia and research development only. IPD requests may also be subjected to SickKids' institutional agreements/contracts. IPD mechanism of sharing and types of analysis/data shared will be directed and determined by SickKids' institutional research contracts requirements
Supporting Information: Study Protocol, SAP
Time Frame: 6 months after publication
Access Criteria: Requests for IPD will be reviewed by the study PI and SickKids institute. IPD will be provided to researchers interested in furthering academia and research development only. IPD requests may also be subjected to SickKids' institutional agreements/contracts. IPD mechanism of sharing and types of analysis/data shared will be directed and determined by SickKids' institutional research contracts requirements.